CLINICAL TRIAL: NCT02223897
Title: Umbilical Cord Mesenchymal Stem Cells Transplantation for Treatment of Patients With Ischemic-type Biliary Lesions After Liver Transplantation
Brief Title: Mesenchymal Stem Cells Transplantation for Ischemic-type Biliary Lesions
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Yang Yang (Other)
Responsible Party: Sponsor-Investigator, Yang Yang, Department of Transplantation, Third Affiliated Hospital, Sun Yat-Sen University
Organization: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2014006
Record Dates: First submitted 2014-08-21; First posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Ischemic-type Biliary Lesions
Keywords: Liver transplantation; Biliary complication; mesenchymal stem cells
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional treatment, huc-MSCs (Experimental): Received conventional treatment and huc-MSCs once per week for the first month and once per month for 6 months(9 times in total), at a dose of 1×106 huc-MSCs/kg body weight.
  Interventions: Drug: huc-MSCs
- Conventional plus placebo (Placebo Comparator): Received conventional treatment and 50 ml saline once per week for the first month and once per month for 6 months(9 times in total).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: huc-MSCs — Received conventional treatment and huc-MSCs once per week for the first month and once per month for 6 months(9 times in total), at a dose of 1×106 huc-MSCs/kg body weight.
  Other Names: Umbilical Cord-Derived Mesenchymal Stem Cells
  Arms: Conventional treatment, huc-MSCs
Drug: Placebo — Received conventional treatment and 50 ml saline solution once per week for the first month and once per month for 6 months(9 times in total).
  Other Names: saline solution
  Arms: Conventional plus placebo

SUMMARY:
Ischemic-type biliary lesions (ITBLs) are a major cause of graft loss and mortality after orthotopic liver transplantation (OLT). For now, there are still lacking effective treatment for ITBLs. The purpose of this study is to confirm whether human umbilical cord mesenchymal stem cells are effective in the treatment,or prevention of Ischemic-type Biliary Lesions after liver transplantation.

DETAILED DESCRIPTION:
Advances in organ preservation techniques, immunosuppressive regimens, and surgical techniques have resulted in reduced rates of infection, acute rejection and vascular complications after orthotopic liver transplantation (OLT). However, ischemic-type biliary lesions (ITBLs) are still one of the most serious complications after OLT, with a usual reported incidence of 5-15%, and an incidence of up to 26% in some studies. 46% patients with ITBLs require re-transplantation after 2 years of OLT.

Mesenchymal stem cells (MSCs),a kind of pluripotent stem cells,can differentiate into vascular endothelial cells, which participate in angiogenesis in ischemic tissue. MSCs can also stimulate the proliferation and migration of mature endothelial cells via paracrine.Furthermore, MSCs secret a variety of cytokines and growth factors, such as vascular endothelial growth factor, human basic fibroblast growth factor, hepatocyte growth factor, interleukin-1 and interleukin-8, etc., which also induce angiogenesis.

Participants in the study will be randomly assigned to one of two treatment arms:

* Arm A: Participants will receive 6 months of standard regular treatment for ITBLs plus huc-MSCs treatment.
* Arm B: Participants will receive 6 months of standard regular treatment for ITBLs plus placebo.

huc-MSCs will be prepared according to standard procedures and is collected in plastic bags containing anti coagulant. MSCs are given via i.v. After huc-MSCs transfusion, patients are followed up once per week(in the first months,<1M),once per 2 week(1-3M)and once per month(3-6M), and the evaluation of liver function and biliary blood supply was performed.

ELIGIBILITY:
Inclusion Criteria:

* benign end-stage liver disease patients with liver transplantation.
* ages of 18 and 60 years.
* first liver transplant.
* gamma-glutamyltransferase > 300 U/L for 2 weeks, and there was no or low enhancement of the wall of the hilar bile duct in arterial phase via contrast-enhanced ultrasonography.
* Written informed consent.

Exclusion Criteria:

* second or combined organ transplant recipient.
* vital organs failure (Cardiac, Renal or Respiratory, et al).
* clinically active bacterial, fungal, viral or parasitic infection.
* other candidates who are judged to be not applicable to this study by investigators.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2014-07; Primary Completion 2017-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
The incidence of ITBLs | 18 months

SECONDARY OUTCOMES:
Changes in biliary enzymology | 18 months
Biliary blood supply | 18 months
  Biliary blood supply indicated by contrast-enhanced ultrasound.

OTHER OUTCOMES:
life quality | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Yang Yang, MD, Study Chair — Third Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong, China